CLINICAL TRIAL: NCT02203604
Title: A Phase II Single Arm Study of High-Dose IL-2 and Ipilimumab in Patients With Unresectable Stage III and Stage IV Melanoma
Brief Title: High-Dose Aldesleukin and Ipilimumab in Treating Patients With Stage III-IV Melanoma That Cannot Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient rate of accrual
Sponsor: CINJRegulatory (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor-Investigator, CINJRegulatory, CINJ Clinical Trial Administrator, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 091309; NCI-2014-01306 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CA184-084; Pro20140000135 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH); Pro20140000135 (Other: IRB number)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2023-06-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Recurrent Melanoma; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interleukin-2; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (aldesleukin, ipilimumab) (Experimental): INDUCTION: Patients receive ipilimumab IV over 90 minutes on days 1, 22, 43, and 64 and high-dose aldesleukin IV on days 22-26 and 43-47.
  MAINTENANCE: Beginning on weeks 24, patients without disease progression or unacceptable toxicity receive ipilimumab IV over 90 minutes once every 12 weeks for up to 24 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: aldesleukin; Biological: ipilimumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: aldesleukin — Given IV
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Biological: ipilimumab — Given IV
  Other Names: anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody; MDX-010; MDX-CTLA-4; monoclonal antibody CTLA-4
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well high-dose aldesleukin and ipilimumab works in treating patients with stage III-IV melanoma that cannot be removed by surgery. Biological therapies, such as aldesleukin, may stimulate or suppress the immune system in different ways and stop tumor cells from growing. Monoclonal antibodies, such as ipilimumab, interfere with the ability of tumor cells to grow and spread. Giving high-dose aldesleukin together with ipilimumab may work better in treating patients with melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The best overall response rate within the first 24 weeks of combination interleukin (IL)-2 (aldesleukin) and ipilimumab using the immune-related response criteria.

SECONDARY OBJECTIVES:

I. Best overall response (BOR). II. Progression-free survival (PFS). III. Disease control rate (DCR). IV. Overall survival. V. To collect data on the safety and feasibility of combined high-dose IL-2 and ipilimumab.

VI. To evaluate the cluster of differentiation (CD)4+ and CD8+ T cell response in the tumor microenvironment and peripheral blood of patients treated on this study.

OUTLINE:

INDUCTION: Patients receive ipilimumab intravenously (IV) over 90 minutes on days 1, 22, 43, and 64 and high-dose aldesleukin IV on days 22-26 and 43-47.

MAINTENANCE: Beginning on weeks 24, patients without disease progression or unacceptable toxicity receive ipilimumab IV over 90 minutes once every 12 weeks for up to 24 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Histologic or cytologic diagnosis of cutaneous melanoma that is considered unresectable (stage III) or metastatic (stage IV); ocular and mucosal melanoma is excluded
* White blood cell (WBC) >= 2000/uL
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets >= 75 x 10^3/uL
* Hemoglobin >= 9 g/dL (>= 80 g/L; may be transfused)
* Creatinine =< 2.0 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN for patients without liver metastasis, =< 5 times for patients with liver metastases
* Bilirubin =< 2.0 x ULN, (except patients with Gilbert's syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* No known active or chronic infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; testing is not required unless clinically suspected
* Performance status (Eastern Cooperative Oncology Group [ECOG] 0-1)
* Patients must have a life expectancy of greater than three months at the start of the trial
* Patients must have a brain magnetic resonance imaging (MRI) that is free of active metastases; metastases that have been treated with radiation or surgical resection, are stable for at least 4 weeks and do not require steroids are eligible
* Patients may have received treatment of completely resected early stage melanoma, comprising interferon, radiation treatment, or experimental vaccine therapy, and in the metastatic setting patient can have had treatment such as chemotherapy, immunotherapy (except prior treatment with ipilimumab and IL-2), and other experimental agent which was completed 4 weeks prior to enrollment
* Normal cardiac stress test for patients over 50 years of age
* Forced expiratory volume in 1 second (FEV1) > 65% of prediction for those patients with extensive pulmonary metastases or chronic pulmonary disease history
* Forced vital capacity (FVC) > 65% of prediction for those patients with extensive pulmonary metastases or chronic pulmonary disease history
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized; in general, the decision for appropriate methods to prevent pregnancy should be determined by discussions between the investigator and the study subject; WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal; post-menopause is defined as:

  * Amenorrhea >= 12 consecutive months without another cause, or
  * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level >= 35 mIU/mL
  * Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential
  * WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours before the start of ipilimumab
  * Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study (and for up to 26 weeks after the last dose of investigational product) in such a manner that the risk of pregnancy is minimized

Exclusion Criteria:

* Any other malignancy form which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix
* Patients with primary ocular or mucosal melanoma are excluded
* Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre syndrome and Myasthenia Gravis)
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea
* Patients with underlying heart conditions who are deemed ineligible for surgery by cardiology consult; patients with reversible ischemic changes on cardiac stress test
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab)
* A history of prior treatment with IL-2, ipilimumab or prior cytotoxic T-lymphocyte antigen 4 (CTLA4) inhibitor or agonist
* Concomitant therapy with any of the following: interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids
* Women of childbearing potential (WOCBP), who:

  * Are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 8 weeks after cessation of study drug, or
  * Have a positive pregnancy test at baseline, or
  * Are pregnant or breastfeeding
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Kaufman, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (6):
- United States (6):
  - Loyola University Medical Center, Maywood, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silk AW, Kaufman HL, Curti B, Mehnert JM, Margolin K, McDermott D, Clark J, Newman J, Bommareddy PK, Denzin L, Najmi S, Haider A, Shih W, Kane MP, Zloza A. High-Dose Ipilimumab and High-Dose Interleukin-2 for Patients With Advanced Melanoma. Front Oncol. 2020 Jan 10;9:1483. doi: 10.3389/fonc.2019.01483. eCollection 2019. PMID 31998643

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Aldesleukin, Ipilimumab): INDUCTION: Patients receive ipilimumab IV over 90 minutes on days 1, 22, 43, and 64 and high-dose aldesleukin IV on days 22-26 and 43-47.
  MAINTENANCE: Beginning on weeks 24, patients without disease progression or unacceptable toxicity receive ipilimumab IV over 90 minutes once every 12 weeks for up to 24 weeks in the absence of disease progression or unacceptable toxicity.
  aldesleukin: Given IV
  ipilimumab: Given IV
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Aldesleukin, Ipilimumab)
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Aldesleukin, Ipilimumab)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate as Determined by mWHO Criteria
Description: Defined as the ratio of the number of participants whose number of participants whose best response is a complete response or partial response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Objective Response Rate as Determined by mWHO Criteria: Defined as the ratio of the number of participants whose number of participants whose best response is a complete response or partial response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  Up to 24 weeks
Arm/Group | Objective Response Rate as Determined by mWHO Criteria
Number analyzed (Participants) | 9
Participants | 1

2. Secondary Outcome: Number of Participants With Adverse Events, Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The number of participants with adverse in each classification of severity and relationship to treatment will be reported.
Time Frame: Up to 60 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Aldesleukin, Ipilimumab)
Number analyzed (Participants) | 9
participants | 7

3. Secondary Outcome: Overall Survival
Description: number of until death from any cause after the start of treatment
Time Frame: Time from the date of registration to the date of death from any cause, assessed up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Aldesleukin, Ipilimumab)
Number analyzed (Participants) | 9
Participants | 5

4. Secondary Outcome: Count of Participants With Increased Effector CD8+ T Cells
Description: Count of participants from the date of diagnosis or the start of treatment.
Time Frame: Time from the date of registration until the date of documented disease progression or death, assessed up to up to 104 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Aldesleukin, Ipilimumab)
Number analyzed (Participants) | 9
Participants | 4

5. Secondary Outcome: Best Overall Response, Defined as the Best Response Across All Time Points
Description: Best overall response was defined as participants who achieved a complete or partial overall response as assessed by the Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions
Time Frame: After the first 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Objective Response Rate as Determined by mWHO Criteria: Defined as the ratio of the number of participants whose best response is a complete response or partial response divided by the total number of participants enrolled who have baseline and post-treatment assessments.
  Up to 24 weeks
Arm/Group | Objective Response Rate as Determined by mWHO Criteria
Number analyzed (Participants) | 9
Participants | 1

6. Secondary Outcome: Count of Participants With Increased Effector CD8+ T Cells - Frequency of Effector CD8+ T Cells
Description: Treatment effect for each patient will be measured as paired differences between pre and post measurements of these parameters at various times. Transformation of the data will be performed if appropriate, e.g. log transformation, and hence treatment effect will be expressed on a log scale. Data relating to immune response will be presented as descriptive summary statistics (such as mean, standard error and 90% confidence intervals [CI]).
  The purity of the CD8+ T cells can then be measured via flow cytometry next the cells are counted and categorized.
Time Frame: Up to 104 weeks
Population: Data was not collected.
Arm/Group | Treatment (Aldesleukin, Ipilimumab)
Number analyzed (Participants) | 0

7. Secondary Outcome: Frequency of CD4+FoxP3+ Regulatory T Cells
Description: Treatment effect for each patient will be measured as paired differences between pre and post measurements of these parameters at various times. Transformation of the data will be performed if appropriate, e.g. log transformation, and hence treatment effect will be expressed on a log scale. Data relating to immune response will be presented as descriptive summary statistics (such as mean, standard error and 90% CI).Using flow cytometry.
Time Frame: Up to 104 weeks
Population: Data was not collected.
Arm/Group | Treatment (Aldesleukin, Ipilimumab)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of three years.
Arm/Group | Treatment (Aldesleukin, Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Aldesleukin, Ipilimumab) (N=9)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Aldesleukin, Ipilimumab) (N=9)
Fatigue (General disorders) | 2
Fever (General disorders) | 2
Chills (General disorders) | 1
Infusion related reaction (General disorders) | 1
Localized edema (General disorders) | 1
Pain (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash pustular (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
External ear inflammation (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Scleral disorder (Eye disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
The trial was closed early due to slow accrual. Early termination lead to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: SAP Protocol_1 (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT02203604/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: SAP Protocol_2 (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT02203604/Prot_SAP_001.pdf
  • Informed Consent Form (2015-09-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT02203604/ICF_002.pdf